CLINICAL TRIAL: NCT06825546
Title: A Multicenter Study Assessing the Efficacy and Safety of Icaritin in Combination With AG Chemotherapy Versus AG Chemotherapy Alone in Patients With Previously Untreated Advanced Pancreatic Ductal Adenocarcinoma
Brief Title: Icaritin in Combination With AG in Patients With Previously Untreated Advanced Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240721
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-04

CONDITIONS: Advanced Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — icaritin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Icaritin + AG chemotherapy (Experimental): Icaritin soft capsules, 600 mg, taken twice daily, should be swallowed with warm water within 30 minutes after breakfast and dinner. If a patient misses a dose and cannot take it within 2 hours after a meal, they should continue with the next scheduled dose without needing to make up for the missed dose.
  Gemcitabine, 1000 mg/m², is administered on days 1 and 8, followed by a 14-day pause, constituting a 21-day treatment cycle. Nab-paclitaxel, 125 mg/m², is also administered on days 1 and 8, with a 14-day pause, making up a 21-day treatment cycle.
  Interventions: Drug: Icaritin; Drug: AG chemotherapy
- AG chemotherapy (Active Comparator): 1. Gemcitabine (1000 mg/m²) + saline (100 mL), infused intravenously over 30 minutes, followed by a 100 mL saline flush.
  2. Nab-paclitaxel (125 mg/m²) + saline (100 mL), infused intravenously over 30 minutes, followed by a 100 mL saline flush
  Interventions: Drug: AG chemotherapy

INTERVENTIONS:
Drug: Icaritin — Icaritin soft capsules, 600 mg, taken twice daily, should be swallowed with warm water within 30 minutes after breakfast and dinner. If a patient misses a dose and cannot take it within 2 hours after a meal, they should continue with the next scheduled dose without needing to make up for the missed dose.
  Gemcitabine, 1000 mg/m², is administered on days 1 and 8, followed by a 14-day pause, constituting a 21-day treatment cycle. Nab-paclitaxel, 125 mg/m², is also administered on days 1 and 8, with a 14-day pause, making up a 21-day treatment cycle.
  Arms: Icaritin + AG chemotherapy
Drug: AG chemotherapy — Gemcitabine (1000 mg/m²) + saline (100 mL), infused intravenously over 30 minutes, followed by a 100 mL saline flush.
  Nab-paclitaxel (125 mg/m²) + saline (100 mL), infused intravenously over 30 minutes, followed by a 100 mL saline flush

SUMMARY:
Icaritin is a drug that has been approved by the National Medical Products Administration (NMPA) based on a multicenter, randomized, double-blind, parallel-controlled Phase III clinical trial - SNG1705 ICR-1. It is used for patients with unresectable hepatocellular carcinoma who are not suitable for or refuse standard treatment and have not previously received systemic therapy. According to numerous studies, in tumor cells, Icaritin can downregulate the expression of TNF-α, IL-6, PD-L1 and exert anti-tumor effects. At the same time, it regulates the tumor immune microenvironment by reducing the secretion of TNFa and IL-6 as well as inhibiting PD-L1 expression through decreasing MDSC cell proportion. Importantly, Icaritin has excellent safety profile and greatly ensure patients' quality of life clinically. Rare grade 3-4 TRAEs were observed in clinical trials which is uncommon among existing standard drugs. Good safety is a prerequisite for combination therapy; therefore, further exploration of optimal drug combinations is worth considering. Thus,we investigated the efficacy and safety of Icaritin administered in conjunction with AG in patients newly diagnosed with advanced pancreatic ductal adenocarcinoma, compare with AG only.

DETAILED DESCRIPTION:
This study aims to evaluate the superiority of Icaritin soft capsules combined with the AG chemotherapy regimen (including gemcitabine) compared to the AG regimen alone. By modulating the immune microenvironment, the combined therapy is expected to provide synergistic enhancement. This will lay the groundwork and provide data for subsequent large-scale randomized controlled clinical trials, ultimately offering more effective combination therapies for patients with advanced pancreatic cancer and improving survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old (including the cutoff value).
2. patients with histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC) disease from multiple centers including Sir Run Run Shaw Hospital, Zhejiang University School of Medicine (group lead unit).
3. locally advanced or metastatic PDAC according to the 2024 CSCO Guidelines for the Management of Pancreatic Cancer.
4. no prior systemic therapy.
5. presence of measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
6. Eastern Cooperative Oncology Group PS 0 or 1.
7. have a life expectancy of at least 3 months.
8. adequate organ function (absolute neutrophil count ≥1.5×109/L; Platelet count ≥100×109/L; Creatinine <1.5×ULN (upper limit of normal) or creatinine clearance (CRCI) ≥60 ml/min; Albumin ≥30g/L; Total bilirubin <5×ULN; Aspartate aminotransferase (AST) <2.5×ULN; Alanine aminotransferase (ALT) <2.5×ULN (≤5×ULN is acceptable if liver metastasis is present); INR or PT < 1.5×ULN, APTT < 1.5×ULN.
9. in a fertile woman, a negative serum pregnancy test within 7 days before the first trial treatment;
10. willingness to use a highly effective contraceptive method (failure rate < 1.0% per year) from the first study treatment until 24 weeks after completion of the trial treatment, if the woman is fertile or the male participant's partner is fertile.
11. no other serious underlying medical conditions.
12. voluntarily participated in this study and signed informed consent. If the subjects were unable to read and sign the informed consent form due to incapacity or other reasons, their guardians were required to act for them during the informed consent process and sign the informed consent form. If the subjects were unable to read the informed consent form (e.g., illiterate subjects), witnesses were required to witness the informed consent process and sign the informed consent.

Exclusion Criteria:

1. neuroendocrine (carcinoid, islet cell) or pancreatic acinar carcinoma.
2. Patients had moderate to severe ascites (ascites was defined by B-ultrasound).
3. untreated active central nervous system or meningeal metastases.
4. Previous systemic therapies such as targeted therapy, immunotherapy, chemotherapy, and modern Chinese medicine with anti-tumor indications or other treatments such as surgery and particle implantation have been used to treat pancreatic cancer.
5. surgery for any reason (other than diagnostic biopsy), within 4 weeks after the first trial treatment, and/or the subject did not fully recover from surgery within 4 weeks after the first trial treatment.
6. history of RT within 3 months of the first dose of trial treatment. No more than 30% bone marrow irradiation or large field irradiation should be used in the 4 weeks before the first trial treatment.
7. patients with a history of other cancers within the past 2 years.
8. major cardiovascular impairment in the 12 months before the first dose of study drug: such as a history of congestive heart failure higher than NYHA class II, unstable angina, myocardial infarction, or stroke due to cerebrovascular accident, or arrhythmia associated with hemodynamic instability; The corrected QT (QTc) interval was prolonged >480ms.
9. with bleeding or thrombotic diseases or receiving thrombolytic therapy, and coagulopathy; Patients who were deemed by the investigator to be ineligible for participation in the study.
10. clinically significant hemoptysis or tumor bleeding of any cause within 2 weeks before the first dose of study intervention.
11. patients with a history of uncontrolled epilepsy, central nervous system disease, or psychiatric illness, or hypertension The investigator will determine whether clinical severity prevents informed consent from being signed or affects patient adherence to oral medication.
12. had active autoimmune disease requiring systemic therapy within the previous 2 years.
13. may have other comorbidities that are relatively contraindicated in this trial.
14. had a severe allergic reaction to the active ingredient of the trial drug.
15. were pregnant or lactating, or were unwilling to plan pregnancy during the trial.
16. any other medical condition that the investigator considered to interfere with the requirements of the trial in terms of safety or efficacy assessment or adherence to treatment.
17. vulnerable groups except the elderly/illiterate, including people with mental illness, cognitive impairment, critically ill patients, pregnant women, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  The proportion of patients with optimal response achieving complete or partial response

SECONDARY OUTCOMES:
PFS | 2 years
  If the patient has not progressed or died at the last follow-up, the date on which the clinician last confirmed that there was no tumor progression will prevail. For patients who are lost to follow-up, the date when the tumor was last recorded as not progressing will be considered. Patients who have started a new treatment prior to progression will have the date their tumor was last recorded prior to the new treatment.
OS | 2 years
  If the patient is still alive at the last follow-up, the date of the clinician's last confirmation of the patient's survival shall prevail. For patients who were lost to follow-up, the date of last recorded patient survival was considered.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No